CLINICAL TRIAL: NCT02476123
Title: Phase 1 Study of Combination Therapy With Mogamulizumab (KW-0761) and Nivolumab (ONO-4538/BMS-936558) in Subjects With Advanced Solid Tumors
Brief Title: Study of Combination Therapy With Mogamulizumab (KW-0761) and Nivolumab (ONO-4538/BMS-936558) in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0761-013
Record Dates: First submitted 2015-06-10; First posted 2015-06-19 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mogamulizumab+Nivolumab (Experimental): During parts 1 and 2, Mogamulizumab and Nivolumab are administered at appropriate intervals.
  Part 1 (Dose Escalation Part) During Cohort 1 to 2, Mogamulizumab and Nivolumab are administered in combination.
  Part 2 (Expansion Part) Patients will be treated with maximum tolerated dose established in the dose escalation part for each combination.
  Interventions: Biological: Mogamulizumab: KW-0761, Nivolumab: (ONO-4538/BMS-936558)

INTERVENTIONS:
Biological: Mogamulizumab: KW-0761, Nivolumab: (ONO-4538/BMS-936558) — i.v. administration

SUMMARY:
The purpose of this study is to characterize the safety and tolerability and determine the maximum tolerated dose (MTD) or the recommended fixed dose of the combinations of Mogamulizumab and Nivolumab in subjects with locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who voluntarily signed and dated Institutional Review Board approved informed consent form in accordance with regulatory and institutional guidelines.
* Subjects who have progressed or have been intolerant to any standard treatment regimen or refused standard treatment, or for which adequate standard therapy does not exist.
* Subjects who have evaluable lesion per guideline of Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Subjects with life expectancy > 12 weeks.
* Subjects with Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1.
* Potential child-bearing female who has agreed with contraception and not breast-feeding. For male who also has agreed with contraception.
* Subjects who have adequate hematological, renal, hepatic and respiratory functions defined.
* Must agree to present archival tumor tissues to sponsor or be willing to undergo a pre-treatment biopsy.
* Histologically or cytologically confirmed locally advanced or metastatic solid tumors.

Exclusion Criteria:

* Female subjects who are pregnant or breast-feeding.
* Subjects with uncontrolled and significant inter-current illness.
* Subjects with known central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Subjects who have been previously treated with an anti-programmed death 1 (PD-1), anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Subjects who have been previously treated with Mogamulizumab.
* Subjects with any prior Grade ≥ 3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE.
* Subjects with a history of severe hypersensitivity reactions to drugs.
* Subjects who have been received chemotherapies, immunotherapy, biologic or hormonal therapies, another investigational drug, radiation or major surgery for cancer treatment within 28 days or 42 days (for nitrosourea or mitomycin C) prior to Cycle 1 Day 1.
* Subjects who have known active autoimmune disease or syndrome.
* Subjects who have active inflammatory bowel disease, irritable bowel disease, celiac disease, or other serious GI chronic conditions associated with diarrhea.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2015-06; Primary Completion 2018-02-07 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting adverse events | From the first dose of study medications until 90 days after the last dose of study medication
Number of subjects reporting serious adverse events | From the first dose of study medications until 90 days after the last dose of study medication
Percentage of subjects reporting serious adverse events | From the first dose of study medications until 90 days after the last dose of study medication
Percentage of subjects reporting adverse events | From the first dose of study medications until 90 days after the last dose of study medication
Number of subjects experiencing dose-limiting toxicity | For 28 days from the first dose of study medications

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Chiba
  - Tokyo

REFERENCES:
- [Derived] Doi T, Muro K, Ishii H, Kato T, Tsushima T, Takenoyama M, Oizumi S, Gemmoto K, Suna H, Enokitani K, Kawakami T, Nishikawa H, Yamamoto N. A Phase I Study of the Anti-CC Chemokine Receptor 4 Antibody, Mogamulizumab, in Combination with Nivolumab in Patients with Advanced or Metastatic Solid Tumors. Clin Cancer Res. 2019 Nov 15;25(22):6614-6622. doi: 10.1158/1078-0432.CCR-19-1090. Epub 2019 Aug 27. PMID 31455681